CLINICAL TRIAL: NCT05849792
Title: Internet-based Physical Activities Randomized Controlled Trial in Patients With Mild/Moderate Depression: Effects on Psychological and Social Well-being: SONRIE Project
Brief Title: Internet-based Physical Activities Randomized Controlled Trial in Mild/Moderate Depression Participants: SONRIE Project
Acronym: SONRIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Junta de Andalucia (Other Government); Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI/0068/2018
Record Dates: First submitted 2023-03-24; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Exercise; Physical Fitness; Depression; Adult ALL; Psychological
Keywords: depression; physical activity; exercise; physical fitness; psychological; Endocannabinoids system
MeSH Terms: conditions — Motor Activity; Depression; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Exercise; Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Group where the participants realize an intervention based on exercise and psychology.
  Interventions: Behavioral: Exercise and psychological intervention
- Control (No Intervention): Group where the subjects do not realize the intervention.

INTERVENTIONS:
Behavioral: Exercise and psychological intervention — Physical Exercise Intervention
  Sixty-minute sessions were delivered via internet, three times per week (1 supervised) over the first four weeks of the COVID-19 home confinement. The intervention was a multicomponent exercise program lead by a specialist in fitness composed of aerobic, resistance, balance, coordination, mobility and stretching exercises. Each multicomponent exercise session consisted of a 10 min warm-up, 40 min of moderate to vigorous intensity physical activity, and 10 min cool down.
  Psychological intervention
  The internet-based-psychological intervention provided to different component of Cognitive Behavioral Therapy (CBT) guided and recorded by a sport neuro-psychologist specialist. The iCBT is based on the protocol for face-to-face CBT for depression. The program consisted of 4 weeks composed of 2 weekly video-guided sessions, with a maximum duration of 30 minutes. iCBT was focused on 4 main axes of action physiological, emotional, behavioral and cognitive.
  Arms: Exercise group

SUMMARY:
The goal of this randomized controlled trial is to determine the effect of an intervention program with physical activity for 12 weeks on depression, social and emotional well-being and quality of life and health in adults with mild and moderate depression. The main questions it aims to answer are:

1. - To determine the association of physical activity levels, sedentary behavior, sleep patterns, physical condition, diet, and general health status with mental and social well-being, and quality of life in a large sample of adult patients diagnosed with mild or moderate depression.
2. - To examine the predictive capacity of physical activity, sedentary behaviors, and physical condition on mild and moderate depressive disorder.
3. - To study the effect of a period without an intervention program with physical activity (8 weeks without exercise intervention) on the variables studied.
4. - To examine the role of the endocannabinoid system on depression as well as its behavior after an intervention program of physical activity.

Participants will be involved in a physical activity intervention program for 12 weeks.

Researchers will compare intervention group and control group to see if an intervention program with physical activity for 12 weeks improve depression, social and emotional well-being and quality of life and health in adults with mild and moderate depression.

DETAILED DESCRIPTION:
One hundred and six eligible participants between 25-65 years old (Spanish higher prevalence of depression in adulthood) diagnosed with mild or moderate depression will be the sample of this project. Participants will be recruited from the Mental Health Unit (UGC Salud Mental), covering different areas of the province of Cadiz (Spain) such as Puerto Real, Chiclana de la Frontera and Vejer de la Frontera. The Mental Health Unit Director from Puerto Real Hospital is a researcher associated with this project who has specific experience with clinical experience. He will be the person in charge for the clinical depression diagnosis. Moreover, participants will perform specific depression tests at the time of recruitment to confirm their clinical status. Individuals who meet the criteria to participate in this study will sign the informed consent previously to their inclusion in this project (see inclusion / exclusion criteria section).

Sample size and statistical power

Sample size determination will be estimated with a 5% type I error (α) and 95% confidence interval establishing a level of precision (d = 0.095) for the hypothesis test to comparing two proportions. The desired sample size will be n = 96 participants and it will be increased by 10% (n = 106) to compensate the possible dropout of participants during the evaluation process of the study. Sample size for the hypothesis test to comparing two means for the intervention study will consider with a significance level alpha of 0.05 and a power of 0.95 (beta = 0.05) and considering the standard deviation for depression variable as 9.36 (Bouldering psychotherapy reduces depressive symptoms even when general physical activity is controlled for: A randomized controlled trial, Heylon, 2018; Mar; 4 (3): e00580). In this way, to detect a minimum mean difference of 8.26 between control and experimental groups for the depression variable, it is estimated that the sample size of each group should be 30 patients. Therefore, a total of 60 participants will be randomly recruited to each group balanced by sex, age and depression clinical severity. It should be taking into account that several simulations to estimate the sample size based on previous studies were performed by STATA statistical software vs. 14.0.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 25-65 years.
* Mild and / or moderate depression diagnosed by Beck Scale.
* Do not have other severe somatic or psychiatric disorders or other diseases that prevents physical activity.
* To be able to communicate with any problem.
* To be able to read and understand the main purpose of the study.
* Informed consent: must be capable and willing to provide consent.

Exclusion Criteria:

* Major depression diagnosed.
* Acute or terminal illness.
* History of cerebral infarction, epilepsy, brain tumor.
* Unstable cardiovascular disease, or other medical conditions.
* Upper or lower extremity fracture in the past 3 months.
* Severe visual or auditory problems.
* Unwillingness to either complete the study requirements or to be randomized into control or training group.
* To be a participant in another research study that may influence the present project.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Depression PRE | month 11-12
  Beck Depression Scale is composed of 21 items that evaluate severity of depression through the assessment of clinical symptoms such as sadness, crying, loss of pleasure, feelings of failure and guilt, thoughts or wishes of suicide, pessimism, etc. That measurements will be measured before the intervention program.
Depression POST | month 18-19
  Beck Depression Scale is composed of 21 items that evaluate severity of depression through the assessment of clinical symptoms such as sadness, crying, loss of pleasure, feelings of failure and guilt, thoughts or wishes of suicide, pessimism, etc. That measurements will be measured immediately after the intervention program.
Depression RET | month 22-23
  Beck Depression Scale is composed of 21 items that evaluate severity of depression through the assessment of clinical symptoms such as sadness, crying, loss of pleasure, feelings of failure and guilt, thoughts or wishes of suicide, pessimism, etc. That measurements will be measured 4 weeks after the intervention program.
Anxiety disorders and stress PRE | month 11-12
  State Anxiety Inventory (STAI), composed of 40 items designed by sentences that describe how the person feels at that moment and how they usually feel, is a measure of trait and state anxiety. That measurements will be measured before the intervention program.
Anxiety disorders and stress POST | month 18-19
  State Anxiety Inventory (STAI), composed of 40 items designed by sentences that describe how the person feels at that moment and how they usually feel, is a measure of trait and state anxiety. That measurements will be measured immediately after the intervention program.
Anxiety disorders and stress RET | month 22-23
  State Anxiety Inventory (STAI), composed of 40 items designed by sentences that describe how the person feels at that moment and how they usually feel, is a measure of trait and state anxiety. That measurements will be measured 4 weeks after the intervention program.
Light physical activity PRE | month 11-12
  Light physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured before the intervention program.
Light physical activity POST | month 18-19
  Light physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured immediately after the intervention program.
Light physical activity RET | month 22-23
  Light physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured 4 weeks after the intervention program.
Moderate physical activity PRE | month 11-12
  Moderate physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured before the intervention program.
Moderate physical activity POST | month 18-19
  Moderate physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured immediately after the intervention program.
Moderate physical activity RET | month 22-23
  Moderate physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured 4 weeks after the intervention program.
Vigorous physical activity PRE | month 11-12
  Vigorous physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured before the intervention program.
Vigorous physical activity POST | month 18-19
  Vigorous physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured immediately after the intervention program.
Vigorous physical activity RET | month 22-23
  Vigorous physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured 4 weeks after the intervention program.
Moderate-Vigorous physical activity PRE | month 11-12
  Vigorous physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured before the intervention program.
Moderate-Vigorous physical activity POST | month 18-19
  Vigorous physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured immediately after the intervention program.
Moderate-Vigorous physical activity RET | month 22-23
  Vigorous physical activity will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured 4 weeks after the intervention program.
Cardiorespiratory fitness PRE | month 11-12
  Measured by the 6-min walking test, which consist of walking the maximum distance possible in 6 minutes. The outcome will be measured in meters. That measurements will be measured before the intervention program.
Cardiorespiratory fitness POST | month 18-19
  Measured by the 6-min walking test, which consist of walking the maximum distance possible in 6 minutes. The outcome will be measured in meters. That measurements will be measured immediately after the intervention program.
Cardiorespiratory fitness RET | month 22-23
  Measured by the 6-min walking test, which consist of walking the maximum distance possible in 6 minutes. The outcome will be measured in meters. That measurements will be measured 4 weeks after the intervention program.
30-s chair stand PRE | month 11-12
  This test consists of getting up and sitting down in a chair as many times as possible in 30 seconds. It measures the ability to get up and sit down in a chair and the result obtained is measured in repetitions. That measurements will be measured before the intervention program.
30-s chair stand POST | month 18-19
  This test consists of getting up and sitting down in a chair as many times as possible in 30 seconds. It measures the ability to get up and sit down in a chair and the result obtained is measured in repetitions. That measurements will be measured immediately after the intervention program.
30-s chair stand RET | month 22-23
  This test consists of getting up and sitting down in a chair as many times as possible in 30 seconds. It measures the ability to get up and sit down in a chair and the result obtained is measured in repetitions. That measurements will be measured 4 weeks after the intervention program.
Chair sit and reach PRE | month 11-12
  The subject is seated on a chair, with one leg extended (the one corresponding to the dominant side). In this position he should try to reach the balls of his feet with his hands without bending the knee. With a tape measure we measure the distance between the tips of the fingers and the tips of the feet. If it does not arrive, the value will be negative. If the value arrives, it will be positive. The flexibility of the lower back, hip extensors and knee flexors is evaluated and the result obtained is measured un centimeters. That measurements will be measured before the intervention program.
Chair sit and reach POST | month 18-19
  The subject is seated on a chair, with one leg extended (the one corresponding to the dominant side). In this position he should try to reach the balls of his feet with his hands without bending the knee. With a tape measure we measure the distance between the tips of the fingers and the tips of the feet. If it does not arrive, the value will be negative. If the value arrives, it will be positive. The flexibility of the lower back, hip extensors and knee flexors is evaluated and the result obtained is measured un centimeters. That measurements will be measured immediately after the intervention program.
Chair sit and reach RET | month 22-23
  The subject is seated on a chair, with one leg extended (the one corresponding to the dominant side). In this position he should try to reach the balls of his feet with his hands without bending the knee. With a tape measure we measure the distance between the tips of the fingers and the tips of the feet. If it does not arrive, the value will be negative. If the value arrives, it will be positive. The flexibility of the lower back, hip extensors and knee flexors is evaluated and the result obtained is measured un centimeters. That measurements will be measured 4 weeks after the intervention program.
Back scratch PRE | month 11-12
  The subject will begin the test in anatomical position, then we will tell him to flex one elbow and raise it behind his head towards his back, the next thing he has to do is bring his opposite arm behind his back and try to touch his middle fingers . It can happen that the fingers touch hearts and it would be zero, if they do not touch we measure with a ruler and it would be negative and if it exceeds we measure positive. It is not allowed under any circumstances to hold the fingers. The arm that goes up is the one that is measured. The flexibility of the upper body is evaluated, specifically of the shoulders and the result obtained is measured in centimeters. That measurements will be measured before the intervention program.
Back scratch POST | month 18-19
  The subject will begin the test in anatomical position, then we will tell him to flex one elbow and raise it behind his head towards his back, the next thing he has to do is bring his opposite arm behind his back and try to touch his middle fingers . It can happen that the fingers touch hearts and it would be zero, if they do not touch we measure with a ruler and it would be negative and if it exceeds we measure positive. It is not allowed under any circumstances to hold the fingers. The arm that goes up is the one that is measured. The flexibility of the upper body is evaluated, specifically of the shoulders and the result obtained is measured in centimeters. That measurements will be measured immediately after the intervention program.
Back scratch RET | month 22-23
  The subject will begin the test in anatomical position, then we will tell him to flex one elbow and raise it behind his head towards his back, the next thing he has to do is bring his opposite arm behind his back and try to touch his middle fingers . It can happen that the fingers touch hearts and it would be zero, if they do not touch we measure with a ruler and it would be negative and if it exceeds we measure positive. It is not allowed under any circumstances to hold the fingers. The arm that goes up is the one that is measured. The flexibility of the upper body is evaluated, specifically of the shoulders and the result obtained is measured in centimeters. That measurements will be measured 4 weeks after the intervention program.
Blind flamingo PRE | month 11-12
  Starting from a standing position, bipedalism, and closed-eyes bring the arms bent to the waist. One leg is raised and we put the big toe of the foot that we have flexed in contact with the ankle of the opposite leg. We will be measuring the leg that is in support with the ground. You have to try to be 60 seconds without falling or losing balance. It will be considered imbalance: removing the hands from their position, removing the contact of the big toe with the ankle, moving the foot that I have in contact with the ground. The static balance of the leg in contact with the ground is evaluated and the result obtained is measured in seconds. That measurements will be measured before the intervention program.
Blind flamingo POST | month 18-19
  Starting from a standing position, bipedalism, and closed-eyes bring the arms bent to the waist. One leg is raised and we put the big toe of the foot that we have flexed in contact with the ankle of the opposite leg. We will be measuring the leg that is in support with the ground. You have to try to be 60 seconds without falling or losing balance. It will be considered imbalance: removing the hands from their position, removing the contact of the big toe with the ankle, moving the foot that I have in contact with the ground. The static balance of the leg in contact with the ground is evaluated and the result obtained is measured in seconds. That measurements will be measured immediately after the intervention program.
Blind flamingo RET | month 22-23
  Starting from a standing position, bipedalism, and closed-eyes bring the arms bent to the waist. One leg is raised and we put the big toe of the foot that we have flexed in contact with the ankle of the opposite leg. We will be measuring the leg that is in support with the ground. You have to try to be 60 seconds without falling or losing balance. It will be considered imbalance: removing the hands from their position, removing the contact of the big toe with the ankle, moving the foot that I have in contact with the ground. The static balance of the leg in contact with the ground is evaluated and the result obtained is measured in seconds. That measurements will be measured 4 weeks after the intervention program.
8 ft. up and go PRE | month 11-12
  It is executed with the participant seated in a chair against the wall, the performer, with his back touching the back of the chair. A cone will be placed at a distance of 2.45m (8 feet) and the test consists of getting up, going around the cone and sitting down in the shortest possible time, without there being a flight phase, that is, you cannot run. Stop the timer when your back touches the back of the chair. It doesn't matter which way you turn the cone. To get up, it is important not to rest your hands on your thighs, normally you are told to cross your arms. Dynamic balance, agility and coordination are evaluated and the result obtained is measured in seconds. That measurements will be measured before the intervention program.
8 ft. up and go POST | month 18-19
  It is executed with the participant seated in a chair against the wall, the performer, with his back touching the back of the chair. A cone will be placed at a distance of 2.45m (8 feet) and the test consists of getting up, going around the cone and sitting down in the shortest possible time, without there being a flight phase, that is, you cannot run. Stop the timer when your back touches the back of the chair. It doesn't matter which way you turn the cone. To get up, it is important not to rest your hands on your thighs, normally you are told to cross your arms. Dynamic balance, agility and coordination are evaluated and the result obtained is measured in seconds. That measurements will be measured immediately after the intervention program.
8 ft. up and go RET | month 22-23
  It is executed with the participant seated in a chair against the wall, the performer, with his back touching the back of the chair. A cone will be placed at a distance of 2.45m (8 feet) and the test consists of getting up, going around the cone and sitting down in the shortest possible time, without there being a flight phase, that is, you cannot run. Stop the timer when your back touches the back of the chair. It doesn't matter which way you turn the cone. To get up, it is important not to rest your hands on your thighs, normally you are told to cross your arms. Dynamic balance, agility and coordination are evaluated and the result obtained is measured in seconds. That measurements will be measured 4 weeks after the intervention program.
Handgrip strength PRE | month 11-12
  This test, also known as a hand grip test, is performed with a dynamometer, which comes in two types, manual and electronic. It measures the force in kilograms, we need to regulate the length of the grip, but it has been shown that there is an optimal grip for men and for women and children. For men it is 5.5 cm. The measurement will be carried out alternately in each hand and a total of two measurements in each hand. Looking straight ahead and there can be no wrist movement, the subject will be told to hold the force for about 3 seconds. The factor that this test evaluates is the isometric strength of the hand and forearm and the result obtained is measured in kilograms. That measurements will be measured before the intervention program.
Handgrip strength POST | month 18-19
  This test, also known as a hand grip test, is performed with a dynamometer, which comes in two types, manual and electronic. It measures the force in kilograms, we need to regulate the length of the grip, but it has been shown that there is an optimal grip for men and for women and children. For men it is 5.5 cm. The measurement will be carried out alternately in each hand and a total of two measurements in each hand. Looking straight ahead and there can be no wrist movement, the subject will be told to hold the force for about 3 seconds. The factor that this test evaluates is the isometric strength of the hand and forearm and the result obtained is measured in kilograms. That measurements will be measured immediately after the intervention program.
Handgrip strength RET | month 22-23
  This test, also known as a hand grip test, is performed with a dynamometer, which comes in two types, manual and electronic. It measures the force in kilograms, we need to regulate the length of the grip, but it has been shown that there is an optimal grip for men and for women and children. For men it is 5.5 cm. The measurement will be carried out alternately in each hand and a total of two measurements in each hand. Looking straight ahead and there can be no wrist movement, the subject will be told to hold the force for about 3 seconds. The factor that this test evaluates is the isometric strength of the hand and forearm and the result obtained is measured in kilograms. That measurements will be measured 4 weeks after the intervention program.
Anandamine (AEA) PRE | month 11-12
  Anandamine (AEA) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured before the intervention program.
Anandamine (AEA) POST | month 18-19
  Anandamine (AEA) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured immediately after the intervention program.
Anandamine (AEA) RET | month 22-23
  Anandamine (AEA) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured 4 weeks after the intervention program.
2-araquinodilglicerol (2-AG) PRE | month 11-12
  2-araquinodilglicerol (2-AG) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured before the intervention program.
2-araquinodilglicerol (2-AG) POST | month 18-19
  2-araquinodilglicerol (2-AG) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured immediately after the intervention program.
2-araquinodilglicerol (2-AG) RET | month 22-23
  2-araquinodilglicerol (2-AG) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured 4 weeks after the intervention program.
N-palmitoylethanolamide (PEA) PRE | month 11-12
  N-palmitoylethanolamide (PEA) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured before the intervention program.
N-palmitoylethanolamide (PEA) POST | month 18-19
  N-palmitoylethanolamide (PEA) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured immediately after the intervention program.
N-palmitoylethanolamide (PEA) RET | month 22-23
  N-palmitoylethanolamide (PEA) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured 4 weeks after the intervention program.
N-oleylethanolamine (OEA) PRE | month 11-12
  N-oleylethanolamine (OEA) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured before the intervention program.
N-oleylethanolamine (OEA) POST | month 18-19
  N-oleylethanolamine (OEA) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured immediately after the intervention program.
N-oleylethanolamine (OEA) RET | month 22-23
  N-oleylethanolamine (OEA) will be quantified by isotopic dilution, liquid chromatography/ electrospray ionization tandem mass spectrometry (LC-ESI-MS). That measurements will be measured 4 weeks after the intervention program.
Brain-derived neurotrophic factor PRE | month 11-12
  It will be analysed in serum by using indirect enzyme-linked immunosorbent assay (ELISA Kit, Chemicon, Temecula, CA, USA) of RAyBio Human BDNF (RAFER). That measurements will be measured before the intervention program.
Brain-derived neurotrophic factor POST | month 18-19
  It will be analysed in serum by using indirect enzyme-linked immunosorbent assay (ELISA Kit, Chemicon, Temecula, CA, USA) of RAyBio Human BDNF (RAFER). That measurements will be measured immediately after the intervention program.
Brain-derived neurotrophic factor RET | month 22-23
  It will be analysed in serum by using indirect enzyme-linked immunosorbent assay (ELISA Kit, Chemicon, Temecula, CA, USA) of RAyBio Human BDNF (RAFER). That measurements will be measured 4 weeks after the intervention program.

SECONDARY OUTCOMES:
Ryff's Psychological Well-Being Scale (42-item) PRE | month 11-12
  Ryff's Psychological Well-Being Scale, evaluates optimal psychological functioning and experience in life. It is composed of 29 items grouped in 6 core dimensions: self-acceptance, positive relationships, autonomy, environmental control, purpose in life, and personal growth. The Ryff's Scale can obtain values from 42 to 294. That measurements will be measured before the intervention program.
Ryff's Psychological Well-Being Scale (42-item) POST | month 18-19
  Ryff's Psychological Well-Being Scale, evaluates optimal psychological functioning and experience in life. It is composed of 29 items grouped in 6 core dimensions: self-acceptance, positive relationships, autonomy, environmental control, purpose in life, and personal growth. The Ryff's Scale can obtain values from 42 to 294. That measurements will be measured immediately after the intervention program.
Ryff's Psychological Well-Being Scale (42-item) RET | month 22-23
  Ryff's Psychological Well-Being Scale, evaluates optimal psychological functioning and experience in life. It is composed of 29 items grouped in 6 core dimensions: self-acceptance, positive relationships, autonomy, environmental control, purpose in life, and personal growth. The Ryff's Scale can obtain values from 42 to 294, being 42 the worst score. That measurements will be measured 4 weeks after the intervention program.
The SF-36 Health Questionnaire PRE | month 11-12
  The SF-36 Health Questionnaire is made up of 36 questions (items) that assess both positive and negative states of health. The 36 items of the instrument cover the following scales: Physical function, Physical role, Bodily pain, General health, Vitality, Social function, Emotional role, and Mental health. The SF-36 can obtain values from 0 to 100, being 0 the worst score. That measurements will be measured before the intervention program.
The SF-36 Health Questionnaire POST | month 18-19
  The SF-36 Health Questionnaire is made up of 36 questions (items) that assess both positive and negative states of health. The 36 items of the instrument cover the following scales: Physical function, Physical role, Bodily pain, General health, Vitality, Social function, Emotional role, and Mental health. The SF-36 can obtain values from 0 to 100, being 0 the worst score. That measurements will be measured immediately after the intervention program.
The SF-36 Health Questionnaire RET | month 22-23
  The SF-36 Health Questionnaire is made up of 36 questions (items) that assess both positive and negative states of health. The 36 items of the instrument cover the following scales: Physical function, Physical role, Bodily pain, General health, Vitality, Social function, Emotional role, and Mental health. The SF-36 can obtain values from 0 to 100, being 0 the worst score. That measurements will be measured 4 weeks after the intervention program.
Blood pressure PRE | month 11-12
  Resting blood pressure (systolic and diastolic) will be measured twice, 2 minutes apart, after 5 minutes at rest, units will be mmHg (M6 upper arm blood pressure monitor Omron, Omron Health Care Europe B.V. Hoolddorp, The Netherlands). That measurements will be measured before the intervention program.
Blood pressure POST | month 18-19
  Resting blood pressure (systolic and diastolic) will be measured twice, 2 minutes apart, after 5 minutes at rest, units will be mmHg (M6 upper arm blood pressure monitor Omron, Omron Health Care Europe B.V. Hoolddorp, The Netherlands). That measurements will be measured immediately after the intervention program.
Blood pressure RET | month 22-23
  Resting blood pressure (systolic and diastolic) will be measured twice, 2 minutes apart, after 5 minutes at rest, units will be mmHg (M6 upper arm blood pressure monitor Omron, Omron Health Care Europe B.V. Hoolddorp, The Netherlands). That measurements will be measured 4 weeks after the intervention program.
Heart rate PRE | month 11-12
  Heart rate will be measured twice, 2 minutes apart, after 5 minutes at rest, units will be bpm (beats per minute) (M6 upper arm blood pressure monitor Omron, Omron Health Care Europe B.V. Hoolddorp, The Netherlands). That measurements will be measured before the intervention program.
Heart rate POST | month 18-19
  Heart rate will be measured twice, 2 minutes apart, after 5 minutes at rest, units will be bpm (beats per minute) (M6 upper arm blood pressure monitor Omron, Omron Health Care Europe B.V. Hoolddorp, The Netherlands). That measurements will be measured immediately after the intervention program.
Heart rate RET | month 22-23
  Heart rate will be measured twice, 2 minutes apart, after 5 minutes at rest, units will be bpm (beats per minute) (M6 upper arm blood pressure monitor Omron, Omron Health Care Europe B.V. Hoolddorp, The Netherlands). That measurements will be measured 4 weeks after the intervention program.
Weight PRE | month 11-12
  Weight will be assessed in accordance with the ISAK guidelines with a Tanita MC-780 MA, 8 electrodes following the standardized protocol. That measurements will be measured before the intervention program.
Weight POST | month 18-19
  Weight will be assessed in accordance with the ISAK guidelines with a Tanita MC-780 MA, 8 electrodes following the standardized protocol. That measurements will be measured immediately after the intervention program.
Weight RET | month 22-23
  Weight will be assessed in accordance with the ISAK guidelines with a Tanita MC-780 MA, 8 electrodes following the standardized protocol. That measurements will be measured 4 weeks after the intervention program.
Height PRE | month 11-12
  Height will be assessed in accordance with the ISAK guidelines with a stadiometer SECA 217 following the standardized protocol. That measurements will be measured before the intervention program.
Height POST | month 18-19
  Height will be assessed in accordance with the ISAK guidelines with a stadiometer SECA 217 following the standardized protocol. That measurements will be measured immediately after the intervention program.
Height RET | month 22-23
  Height will be assessed in accordance with the ISAK guidelines with a stadiometer SECA 217 following the standardized protocol. That measurements will be measured 4 weeks after the intervention program.
Waist circumference PRE | month 11-12
  Waist circumference will be assessed in accordance with the ISAK guidelines with a circumference tape SECA following the standardized protocol. That measurements will be measured before the intervention program.
Waist circumference POST | month 18-19
  Waist circumference will be assessed in accordance with the ISAK guidelines with a circumference tape SECA following the standardized protocol. That measurements will be measured immediately after the intervention program.
Waist circumference RET | month 22-23
  Waist circumference will be assessed in accordance with the ISAK guidelines with a circumference tape SECA following the standardized protocol. That measurements will be measured 4 weeks after the intervention program.
Fat mass PRE | month 11-12
  Fat mass will be assessed in accordance with the ISAK guidelines with a Tanita MC-780 MA, 8 electrodes following the standardized protocol. That measurements will be measured before the intervention program.
Fat mass POST | month 18-19
  Fat mass will be assessed in accordance with the ISAK guidelines with a Tanita MC-780 MA, 8 electrodes following the standardized protocol. That measurements will be measured immediately after the intervention program.
Fat mass RET | month 22-23
  Fat mass will be assessed in accordance with the ISAK guidelines with a Tanita MC-780 MA, 8 electrodes following the standardized protocol. That measurements will be measured 4 weeks after the intervention program.
Sociodemographic characteristics questionnaire PRE | month 11-12
  Age, sex, marital status, educational level, socioeconomic status, family history of depression, self-rated health status, consumption of medicines and other pathologies will be determined by this questionnaires. That measurements will be measured before the intervention program.
Sociodemographic characteristics questionnaire POST | month 18-19
  Age, sex, marital status, educational level, socioeconomic status, family history of depression, self-rated health status, consumption of medicines and other pathologies will be determined by this questionnaires. That measurements will be measured immediately after the intervention program.
Sociodemographic characteristics questionnaire RET | month 22-23
  Age, sex, marital status, educational level, socioeconomic status, family history of depression, self-rated health status, consumption of medicines and other pathologies will be determined by this questionnaires. That measurements will be measured 4 weeks after the intervention program.
Food Frequency Questionnaire (FFQ) PRE | month 11-12
  food frequency questionnaire (FFQ) consists of a finite list of foods and beverages with response categories to indicate usual frequency of consumption over the time period queried. To assess the total diet, the number of foods and beverages queried typically ranges from 80 to 120. That measurements will be measured before the intervention program.
Food Frequency Questionnaire (FFQ) POST | month 18-19
  food frequency questionnaire (FFQ) consists of a finite list of foods and beverages with response categories to indicate usual frequency of consumption over the time period queried. To assess the total diet, the number of foods and beverages queried typically ranges from 80 to 120. That measurements will be measured immediately after the intervention program.
Food Frequency Questionnaire (FFQ) RET | month 22-23
  food frequency questionnaire (FFQ) consists of a finite list of foods and beverages with response categories to indicate usual frequency of consumption over the time period queried. To assess the total diet, the number of foods and beverages queried typically ranges from 80 to 120. That measurements will be measured 4 weeks after the intervention program.
Sleep time PRE | month 11-12
  Sleep time will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured before the intervention program.
Sleep time POST | month 18-19
  Sleep time will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured immediately after the intervention program.
Sleep time RET | month 22-23
  Sleep time will be assessed by accelerometers (Actigraph GT3X, MTI, USA) for seven consecutive days with a minimum of 3 days (1 day from weekend) and at less 8 valid hours/day of data collection. The ActiLife Software version 6.13.3 will be used to manage the data. That measurements will be measured 4 weeks after the intervention program.
The Pittsburg Sleep Quality Index PRE | month 11-12
  The Pittsburg Sleep Quality Index will be administer to assess sleep quality and disturbances over a month time interval. It is self-rated questionnaire composed of 19 items that assess 7 components of sleep, covering subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction. That measurements will be measured before the intervention program.
The Pittsburg Sleep Quality Index POST | month 18-19
  The Pittsburg Sleep Quality Index will be administer to assess sleep quality and disturbances over a month time interval. It is self-rated questionnaire composed of 19 items that assess 7 components of sleep, covering subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction. That measurements will be measured immediately after the intervention program.
The Pittsburg Sleep Quality Index RET | month 22-23
  The Pittsburg Sleep Quality Index will be administer to assess sleep quality and disturbances over a month time interval. It is self-rated questionnaire composed of 19 items that assess 7 components of sleep, covering subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction. That measurements will be measured 4 weeks after the intervention program.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cádiz, Puerto Real, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richter P, Werner J, Heerlein A, Kraus A, Sauer H. On the validity of the Beck Depression Inventory. A review. Psychopathology. 1998;31(3):160-8. doi: 10.1159/000066239. PMID 9636945
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Spielberger CD, Gorsuch RL, L. R. State-trait anxiety inventory. Palo Alto Consult. Psychol. Press 1-23 (1970)
- [Background] Ryff, C. D. Happiness is everything, or is it? Explorations on the meaning of psychological well-being. J. Pers. Soc. Psychol. 57, 1069-1081 (1989)
- [Background] Diaz D, Rodriguez-Carvajal R, Blanco A, Moreno-Jimenez B, Gallardo I, Valle C, van Dierendonck D. [Spanish adaptation of the Psychological Well-Being Scales (PWBS)]. Psicothema. 2006 Aug;18(3):572-7. Spanish. PMID 17296089
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Vilagut G, Ferrer M, Rajmil L, Rebollo P, Permanyer-Miralda G, Quintana JM, Santed R, Valderas JM, Ribera A, Domingo-Salvany A, Alonso J. [The Spanish version of the Short Form 36 Health Survey: a decade of experience and new developments]. Gac Sanit. 2005 Mar-Apr;19(2):135-50. doi: 10.1157/13074369. Spanish. PMID 15860162
- [Background] Pietrobelli A, Rubiano F, St-Onge MP, Heymsfield SB. New bioimpedance analysis system: improved phenotyping with whole-body analysis. Eur J Clin Nutr. 2004 Nov;58(11):1479-84. doi: 10.1038/sj.ejcn.1601993. PMID 15138459
- [Background] Di Marzo V, Matias I. Endocannabinoid control of food intake and energy balance. Nat Neurosci. 2005 May;8(5):585-9. doi: 10.1038/nn1457. PMID 15856067
- [Background] Kroes R, Muller D, Lambe J, Lowik MR, van Klaveren J, Kleiner J, Massey R, Mayer S, Urieta I, Verger P, Visconti A. Assessment of intake from the diet. Food Chem Toxicol. 2002 Feb-Mar;40(2-3):327-85. doi: 10.1016/s0278-6915(01)00113-2. PMID 11893401
- [Background] Martinez-Gonzalez MA, Fernandez-Jarne E, Serrano-Martinez M, Wright M, Gomez-Gracia E. Development of a short dietary intake questionnaire for the quantitative estimation of adherence to a cardioprotective Mediterranean diet. Eur J Clin Nutr. 2004 Nov;58(11):1550-2. doi: 10.1038/sj.ejcn.1602004. PMID 15162136
- [Background] Gonzalez Carrascosa R, Bayo Monto JL, Meneu Barreira T, Garcia Segovia P, Martinez-Monzo J. Design of a self-administered online food frequency questionnaire (FFQ) to assess dietary intake among university population. Nutr Hosp. 2011 Nov-Dec;26(6):1440-6. doi: 10.1590/S0212-16112011000600035. PMID 22411394
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771